CLINICAL TRIAL: NCT01438489
Title: A Phase 2, Randomized Study to Evaluate the Efficacy and Safety of MEDI-546 in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of the Efficacy and Safety of MEDI-546 in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-IA-MEDI-546-1013
Record Dates: First submitted 2011-09-09; First posted 2011-09-22 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: MEDI-546; Anifrolumab; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anifrolumab (MEDI-546) 300 mg (Experimental): Participants will receive 300 milligram (mg) anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
  Interventions: Biological: Anifrolumab 300 mg
- Anifrolumab (MEDI-546) 1000 mg (Experimental): Participants will receive 1000 mg anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
  Interventions: Biological: Anifrolumab 1000 mg
- Matching Placebo (Placebo Comparator): Participants will receive placebo matched to anifrolumab intravenous (IV) infusion every 4 weeks for 48 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Anifrolumab 300 mg — Participants will receive 300 milligram (mg) anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
  Other Names: MEDI-546
  Arms: Anifrolumab (MEDI-546) 300 mg
Biological: Anifrolumab 1000 mg — Participants will receive 1000 mg anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
  Other Names: MEDI-546
  Arms: Anifrolumab (MEDI-546) 1000 mg
Other: Placebo — Participants will receive placebo matched to anifrolumab intravenous (IV) infusion every 4 weeks for 48 weeks.
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MEDI-546 compared to placebo in subjects with chronic, moderately-to-severely active systemic lupus erythematosus (SLE) with an inadequate response to standard of care treatment for SLE.

DETAILED DESCRIPTION:
This is a Phase 2, multinational, multicenter, randomized, double-blind, placebo controlled, parallel-group study to evaluate the efficacy and safety of 2 intravenous (IV) treatment regimens in adult participants with chronic, moderately-to-severely active SLE with an inadequate response to SOC SLE. The investigational product (anifrolumab or placebo) will be administered as a fixed dose every 4 weeks (28 days) for a total of 13 doses.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills at least 4 of the 11 American College of Rheumatology (ACR) criteria for systemic lupus erythematosus (SLE) including a positive antinuclear antibody (ANA) greater than or equal to 1:80 or elevated anti-double-stranded DNA or anti-Smith antibody at screening
* Pediatric or adult SLE with chronic disease activity for greater than or equal to 24 weeks
* Weight greater than or equal to 40 kg
* Currently receiving stable dose of oral prednisone (or equivalent) less than or equal to 40 mg/day and/or antimalarials/immunosuppressives
* Active moderate to severe SLE disease based on SLE disease activity score (SLEDAI) and British Isles Lupus Assessment Group Index (BILAG) and Physicians Global Assessment
* No evidence of cervical malignancy on Pap smear within 2 years of randomization
* Female participants must be willing to avoid pregnancy
* Negative tuberculosis (TB) test or newly positive TB test due to latent TB for which treatment must be initiated at or before randomization.

Exclusion Criteria:

* Active severe SLE-driven renal disease or unstable renal disease prior to screening
* Active severe or unstable neuropsychiatric SLE
* Clinically significant active infection including ongoing and chronic infections
* History of human immunodeficiency virus (HIV)
* Confirmed Positive tests for hepatitis B or positive test for hepatitis C
* History of severe herpes infection such as herpes encephalitis, ophthalmic herpes, disseminated herpes
* Live or attenuated vaccine within 4 weeks prior to screening
* Participants with significant hematologic abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Greth, MD, Study Director — MedImmune LLC
Locations (79):
- United States (30):
  - Research Site, Birmingham, Alabama
  - Research Site, La Jolla, California
  - Research Site, La Palma, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Desert, California
  - Research Site, San Leandro, California
  - Research Site, Upland, California
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Las Cruces, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
- Brazil (2):
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Colombia (5):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Chía
  - Research Site, Medellín
- Czechia (3):
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- India (6):
  - Research Site, Dantoli-Nagpur
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Secunderabad
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, México
  - Research Site, Toluca
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Nadarzyn
  - Research Site, Poznan
- Romania (3):
  - Research Site, Brasov
  - Research Site, Iași
  - Research Site, Târgu Mureş
- South Korea (4):
  - Research Site, Gwangjin-gu
  - Research Site, Gwangju
  - Research Site, Seodaemun-gu
  - Research Site, Suwon
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (7):
  - Research Site, Donetsk
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Ternopil
  - Research Site, Vinnitsya
  - Research Site, Vinnytsia

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Casey KA, Smith MA, Sinibaldi D, Seto NL, Playford MP, Wang X, Carlucci PM, Wang L, Illei G, Yu B, Wang S, Remaley AT, Mehta NN, Kaplan MJ, White WI. Modulation of Cardiometabolic Disease Markers by Type I Interferon Inhibition in Systemic Lupus Erythematosus. Arthritis Rheumatol. 2021 Mar;73(3):459-471. doi: 10.1002/art.41518. Epub 2021 Feb 15. PMID 32909675
- [Derived] Brohawn PZ, Streicher K, Higgs BW, Morehouse C, Liu H, Illei G, Ranade K. Type I interferon gene signature test-low and -high patients with systemic lupus erythematosus have distinct gene expression signatures. Lupus. 2019 Nov;28(13):1524-1533. doi: 10.1177/0961203319885447. Epub 2019 Oct 29. PMID 31660791
- [Derived] Casey KA, Guo X, Smith MA, Wang S, Sinibaldi D, Sanjuan MA, Wang L, Illei GG, White WI. Type I interferon receptor blockade with anifrolumab corrects innate and adaptive immune perturbations of SLE. Lupus Sci Med. 2018 Nov 22;5(1):e000286. doi: 10.1136/lupus-2018-000286. eCollection 2018. PMID 30538817
- [Derived] Morand EF, Trasieva T, Berglind A, Illei GG, Tummala R. Lupus Low Disease Activity State (LLDAS) attainment discriminates responders in a systemic lupus erythematosus trial: post-hoc analysis of the Phase IIb MUSE trial of anifrolumab. Ann Rheum Dis. 2018 May;77(5):706-713. doi: 10.1136/annrheumdis-2017-212504. Epub 2018 Feb 2. PMID 29420200
- [Derived] Furie R, Khamashta M, Merrill JT, Werth VP, Kalunian K, Brohawn P, Illei GG, Drappa J, Wang L, Yoo S; CD1013 Study Investigators. Anifrolumab, an Anti-Interferon-alpha Receptor Monoclonal Antibody, in Moderate-to-Severe Systemic Lupus Erythematosus. Arthritis Rheumatol. 2017 Feb;69(2):376-386. doi: 10.1002/art.39962. PMID 28130918

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 626 participants were screened out of which 319 participants did not meet eligibility criteria and were considered screen failures, and 307 participants were randomized into the study.
Groups:
- Placebo: Participants received placebo matched to anifrolumab intravenous (IV) infusion every 4 weeks for 48 weeks.
- Anifrolumab 300 mg: Participants received 300 milligram (mg) anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
- Anifrolumab 1000 mg: Participants received 1000 mg anifrolumab as an intravenous infusion every 4 weeks for 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Started | 103 | 100 | 104
Completed | 77 | 84 | 85
Not Completed | 26 | 16 | 19
Not completed — Lost to Follow-up | 4 | 2 | 2
Not completed — Withdrawal by Subject | 11 | 3 | 8
Not completed — Death | 0 | 0 | 1
Not completed — Sponsor decision | 4 | 1 | 4
Not completed — Subject choice/Subject moved | 2 | 1 | 1
Not completed — Investigator decision | 0 | 1 | 0
Not completed — AE/SAEs | 2 | 1 | 1
Not completed — Received prohibited medication | 1 | 0 | 0
Not completed — Did not complete all 3 follow-up visits | 2 | 5 | 2
Not completed — Inadequate venous access | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg | Total
Number analyzed (Participants) | 103 | 100 | 104 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (12.9) | 39.3 (12.0) | 40.8 (11.6) | 39.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 94 | 99 | 287
  Male | 9 | 6 | 5 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 0 | 4 | 1 | 5
  Asian | 13 | 3 | 6 | 22
  Black or African American | 12 | 19 | 10 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 41 | 36 | 51 | 128
  Other | 36 | 37 | 36 | 109
  Multiple category checked | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: Participants]
  BRAZIL | 3 | 0 | 0 | 3
  BULGARIA | 3 | 2 | 4 | 9
  COLOMBIA | 16 | 10 | 18 | 44
  CZECH REPUBLIC | 1 | 0 | 2 | 3
  HUNGARY | 2 | 5 | 3 | 10
  INDIA | 2 | 1 | 0 | 3
  MEXICO | 4 | 7 | 5 | 16
  PERU | 15 | 22 | 13 | 50
  POLAND | 11 | 9 | 12 | 32
  ROMANIA | 1 | 0 | 1 | 2
  SOUTH KOREA | 3 | 0 | 3 | 6
  TAIWAN | 7 | 2 | 3 | 12
  UKRAINE | 7 | 4 | 11 | 22
  UNITED STATES OF AMERICA | 28 | 38 | 29 | 95
Baseline weight [Mean (Standard Deviation); unit: kilogram] | 68.08 (18.98) | 69.62 (17.09) | 70.74 (17.29) | 69.48 (17.79)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Systemic Lupus Erythematosus (SLE) Responder Index [SRI (4)] Response With Oral Corticosteroids (OCS) Tapering at Day 169
Description: An SRI (4) responder defined as a participant who had 1) a reduction in baseline Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score of greater than or equal to (>=) 4 points; 2) no worsening of disease from baseline as measured by the Physician Global Assessment (MDGA) (worsening was defined as an increase of >= 0.3 from baseline on a 0 to 3.0 visual analog scale); and 3) no new British Isles Lupus Assessment Group 2004 (BILAG-2004) Index 'A' organ system score and no more than one new or worsening BILAG-2004 Index 'B' organ system score. OCS tapering requires a sustained reduction of OCS from Day 85 through Day 169 [less than 10 milligram per day (mg/day) and less or equal to the dose received on Day 1]. SRI was analyzed by a logistic regression model.
Time Frame: Day 169
Population: The modified Intent-To-Treat (mITT) population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies evaluable participants for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 102 | 99 | 104
Percentage of Participants | 17.6 | 34.3 | 28.8
Statistical Analysis 1: Comparison: Placebo vs Anifrolumab 300 mg; All-comers; Test type: Superiority or Other; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 2.38, 90% CI 2-sided [1.33 to 4.26]
Statistical Analysis 2: Comparison: Placebo vs Anifrolumab 1000 mg; All-comers; Test type: Superiority or Other; p = 0.063, Regression, Logistic; Odds Ratio (OR) = 1.94, 90% CI 2-sided [1.08 to 3.49]

2. Primary Outcome: Percentage of Type I Interferon (IFN) Test High Participants Achieving an Systemic Lupus Erythematosus Responder Index (SRI) (4) Response With Oral Corticosteroids (OCS) Tapering at Day 169
Description: Type I IFN signature in whole blood assessed by using a 4-gene diagnostic test. The blood samples collected were to be used to prospectively identify participants as IFN test-high or test-low. The results of this test were used to stratify participants. An SRI (4) Responder was defined as a participant who had 1) a reduction in baseline SLEDAI-2K disease activity score of >= 4 points; 2) no worsening of disease from baseline as measured by the Physician Global Assessment (MDGA) (worsening was defined as an increase of >= 0.3 from baseline on a 0 to 3.0 visual analog scale); and 3) no new British Isles Lupus Assessment Group 2004 (BILAG-2004) Index A organ system score and no more than one new or worsening BILAG-2004 Index B organ system score. OCS tapering requires a sustained reduction of OCS from Day 85 through Day 169 [less than 10 mg/day and less or equal to the dose received on Day 1]. SRI was analyzed by a logistic regression model.
Time Frame: Day 169
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies evaluable participants for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 76 | 75 | 78
Percentage of Participants | 13.2 | 36 | 28.2
Statistical Analysis 1: Comparison: Placebo vs Anifrolumab 300 mg; High; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 3.55, 90% CI 2-sided [1.72 to 7.32]
Statistical Analysis 2: Comparison: Placebo vs Anifrolumab 1000 mg; High; Test type: Superiority or Other; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 2.65, 90% CI 2-sided [1.27 to 5.53]

3. Secondary Outcome: Percentage of Participants Achieving an Systemic Lupus Erythematosus (SLE) Responder Index [SRI (4)] Response With Oral Corticosteroids (OCS) Tapering at Day 365
Description: An SRI (4) Responder was defined as a participant who had 1) a reduction in baseline SLEDAI-2K disease activity score of >= 4 points; 2) no worsening of disease from baseline as measured by the MDGA (worsening was defined as an increase of >= 0.3 from baseline on a 0 to 3.0 visual analog scale); and 3) no new British Isles Lupus Assessment Group 2004 (BILAG-2004) Index A organ system score and no more than one new or worsening BILAG-2004 Index B organ system score. OCS tapering requires a sustained reduction of OCS from Day 281 through Day 365 (less than 10 mg/day and less or equal to the dose received on Day 1). SRI was analyzed by a logistic regression model.
Time Frame: Day 365
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 102 | 99 | 104
Percentage of Participants | 25.5 | 51.5 | 38.5

4. Secondary Outcome: Percentage of Participants on Oral Corticosteroids (OCS) >=10 mg/Day of Prednisone or Equivalent at Baseline Who Were Able to Taper to Less Than or Equal to (<=) 7.5 mg/Day at Day 365
Description: Participants on OCS >=10 mg/day of prednisone or equivalent at baseline who were able to taper to <= 7.5 mg/day at Day 365 were evaluated.
Time Frame: Day 365
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 64 | 55 | 63
Percentage of Participants | 26.6 | 56.4 | 31.7

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. A serious AE (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly (in offspring of participant). AEs may be treatment emergent (TE) [that is, occurring after initial receipt of investigational product] or non-TE. An AESI is one of scientific and medical concern specific to understanding biologics and requires close monitoring and rapid communication by investigator to sponsor.
Time Frame: Day 1 (Baseline) to Day 422 (End of Study)
Population: The safety population included participants who received any investigational product. Here, "N" signifies evaluable participants for this outcome measure. One participant from Placebo group received Anifrolumab 1000 mg once and hence, included it in the Anifrolumab 1000 mg group.
Measure: Number; unit: Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 101 | 99 | 105
Participants
  TEAEs | 78 | 84 | 90
  TESAEs | 19 | 16 | 18
  AESIs | 12 | 10 | 15

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Investigations Reported as Treatment-Emergent Adverse Events
Description: Any medically significant change in laboratory evaluations were recorded as Treatment emergent adverse events.
Time Frame: Day 1 (Baseline) to Day 422 (End of Study)
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 101 | 99 | 105
Participants
  Neutrophil count increased | 0 | 1 | 3
  Leukocytosis | 0 | 1 | 2
  Leukopenia | 2 | 0 | 3
  Neutropenia | 0 | 0 | 3
  Anaemia | 0 | 0 | 2
  Iron deficiency anaemia | 0 | 1 | 1
  Lymphopenia | 0 | 0 | 2
  Microcytic anaemia | 1 | 0 | 2
  Thrombocytosis | 0 | 1 | 0
  White blood cell count increased | 0 | 0 | 1
  Monocyte count increased | 0 | 0 | 1
  Hypochromic anaemia | 1 | 0 | 0
  Hyperglycaemia | 1 | 3 | 1
  Hypokalaemia | 2 | 3 | 0
  Hepatic enzyme increased | 1 | 0 | 3
  Hypocalcaemia | 0 | 1 | 1
  Lipid metabolism disorder | 0 | 1 | 1
  Alanine aminotransferase increased | 0 | 1 | 1
  Aspartate aminotransferase increased | 0 | 2 | 0
  Blood creatine phosphokinase increased | 0 | 1 | 1
  Hyperlipidaemia | 1 | 0 | 1
  Hypertriglyceridaemia | 2 | 1 | 0
  Hyponatraemia | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0
  Glomerular filtration rate decreased | 0 | 1 | 0
  Transaminases increased | 1 | 0 | 1
  Dyslipidaemia | 1 | 0 | 0
  Alanine aminotransferase abnormal | 1 | 0 | 0
  Aspartate aminotransferase abnormal | 1 | 0 | 0
  Blood triglycerides abnormal | 1 | 0 | 0
  Glomerular filtration rate increased | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Vital Signs Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign parameters are temperature, blood pressure, respiratory rate, heart rate and weight. Vital signs abnormalities were reported as TEAEs.
Time Frame: Day 1 (Baseline) to Day 422 (End of Study)
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 101 | 99 | 105
Participants
  Hypertension | 7 | 3 | 2
  Pyrexia | 5 | 0 | 3
  Blood pressure increased | 0 | 2 | 1
  Blood pressure decreased | 0 | 0 | 1
  Hypotension | 0 | 1 | 0
  Secondary hypertension | 0 | 0 | 1
  Weight increased | 0 | 0 | 1
  Blood pressure abnormal | 1 | 0 | 0
  Chills | 1 | 0 | 0
  Hypertensive emergency | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Any medically significant changes from the screening ECG was recorded as TEAEs. An abnormal ECG findings such as QT prolonged were reported as treatment emergent adverse events.
Time Frame: Day 1 (Baseline) to Day 422 (End of Study)
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 101 | 99 | 105
Participants | 0 | 0 | 2

9. Secondary Outcome: Percentage of SLE Participants With Positive Anti-drug Antibody (ADA)
Description: Anti-drug antibody responses to anifrolumab in serum were evaluated.
Time Frame: Days 1, 85, 141, 169, 253, 337 (Treatment Phase), 365, 396, and 422 (Follow-up Period)
Population: The safety population included participants who received any investigational product. Here, "N" and "n" signifies evaluable participants for this outcome measure and for specified category of the arms respectively. One participant from Placebo group received Anifrolumab 1000 mg once and hence, included it in Anifrolumab 1000 mg group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 101 | 99 | 105
Percentage of Participants
  Day 1 (n=100,98,105) | 1.0 | 1.0 | 1.9
  Day 85 (n=91,93,98) | 1.1 | 0.0 | 0.0
  Day 141 (n=84,94,93) | 2.4 | 0.0 | 2.2
  Day 169 (n=81,89,92) | 2.5 | 0.0 | 1.1
  Day 253 (n=72,86,86) | 0.0 | 1.2 | 0.0
  Day 337 (n=70,87,76) | 0.0 | 1.1 | 0.0
  Day 365 (n=85,96,94) | 0.0 | 1.0 | 1.1
  Day 396 (n=78,88,90) | 0.0 | 2.3 | 0.0
  Day 422 (n=76,86,77) | 1.3 | 5.8 | 0.0
  Any Visit Post Baseline (n= 99,98,102) | 3.0 | 5.1 | 2.0

10. Secondary Outcome: Neutralization Ratio of 21-Gene Type I Interferon (IFN) Signature for Participants With Positive Baseline Pharmacodynamic (PD) Gene Signature
Description: The PD positive and negative gene signature was determined by comparing the expression of type I IFN-inducible genes in a 21-gene panel in study participants relative to pooled normal blood collected from healthy participants.
Time Frame: Days 29, 85, 141, 169, 253, 337 (treatment phase), on Days 365, 396, and 422 (follow up period)
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies evaluable participants for this outcome measure and "n" signifies evaluable participants for the specified category of the arms respectively.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 102 | 99 | 104
Ratio
  Day 29 (n= 68, 66, 73) | -0.753 (44.678) | 70.194 (40.028) | 82.056 (16.108)
  Day 85 (n= 63, 62, 72) | -5.412 (44.354) | 72.639 (34.443) | 79.350 (40.428)
  Day 141 (n= 59, 64, 68) | -25.411 (78.391) | 73.662 (36.684) | 88.569 (10.364)
  Day 169 (n= 56, 60, 66) | -17.122 (67.603) | 77.364 (30.733) | 88.126 (10.278)
  Day 253 (n= 50, 60, 61) | -9.908 (49.826) | 73.972 (41.267) | 86.099 (15.615)
  Day 337 (n= 49, 59, 53) | -13.784 (45.541) | 79.363 (28.803) | 87.811 (8.410)
  Day 365 (n= 58, 66, 68) | -6.428 (50.358) | 72.796 (35.552) | 81.115 (53.121)
  Day 396 (n= 56, 61, 64) | -22.106 (64.529) | 11.510 (56.385) | 72.291 (31.182)
  Day 422 (n= 53, 57, 55) | -31.777 (70.173) | -0.836 (44.596) | 37.532 (66.339)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Anifrolumab at Day 1, 169 and 337
Description: Maximum plasma concentration (Cmax) was defined as the peak plasma level of anifrolumab, derived from plasma concentration -time data.
Time Frame: Pre-infusion and 15 minutes post-infusion on Day 1, 169 and 337
Population: The Pharmacokinetic population included all treated participants with at least 1 Pharmacokinetic assessment. Here, "N" signifies evaluable participants for this outcome measure and "n" signifies evaluable participants for the specified category of the arms respectively.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 98 | 104
micrograms/milliliter (mcg/mL)
  Day 1 (n=98,104) | 82.8 (64.5) [1.33 to 4.26] | 248 (79.9)
  Day 169 (n=86,87) | 110 (63.7) | 375 (137)
  Day 337 (n=83,67) | 127 (64.6) | 439 (140)

12. Secondary Outcome: Accumulation Ratio of Maximum Observed Plasma Concentration (Cmax,AR) of Anifrolumab
Description: Accumulation ratio for maximum plasma concentration (Cmax,AR) of anifrolumab after multiple administration at Day 169 and 337 was calculated.
Time Frame: Pre-infusion and 15 minutes post-infusion on Day 169 and 337
Population: as for outcome 11
Measure: Median (Full Range); unit: Ratio
Arm/Group | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 81 | 86
Ratio
  Day 169 (n=81,86) | 1.36 (63.7) [0.0367 to 3680] | 1.43 (137) [0.211 to 191]
  Day 337 (n=78,66) | 1.56 (64.6) [0.132 to 7050] | 1.76 (140) [0.492 to 240]

13. Secondary Outcome: Trough Concentration (Ctrough) of Anifrolumab at Day 29, 169 and 365
Description: Trough concentration (Ctrough) of anifrolumab at Day 29, 169 and 365 were calculated.
Time Frame: Pre-infusion and 15 minutes post-infusion on Day 29, 169 and 365
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 95 | 99
microgram per milliliter
  Day 29 (n=95,99) | 7.95 (6.17) [0.0367 to 3680] | 46.8 (24.6) [0.211 to 191]
  Day 169 (n=87,87) | 18.4 (12.9) [0.132 to 7050] | 110 (60.5) [0.492 to 240]
  Day 365 (n=83,71) | 23.6 (15.5) | 154 (89.2)

14. Secondary Outcome: Accumulation Ratio of Trough Concentration (Ctrough,AR) of Anifrolumab at Day 169 and 365
Description: Accumulation ratio for trough concentration (Ctrough,AR) of anifrolumab after multiple administration at Day 169 and 365 was calculated.
Time Frame: Pre-infusion and 15 minutes post-infusion on Day 169 and 365
Population: as for outcome 11
Measure: Median (Full Range); unit: Ratio
Arm/Group | Anifrolumab 300 mg | Anifrolumab 1000 mg
Number analyzed (Participants) | 82 | 86
Ratio
  Day 169 (n=82,86) | 2.49 (63.7) [0.0599 to 1250] | 2.29 (137) [0.299 to 30.1]
  Day 365 (n=79,70) | 3.06 (64.6) [0.00816 to 1130] | 3.02 (140) [0.672 to 11.7]

ADVERSE EVENTS:
Time Frame: Day 1 (Baseline) to Day 422 (End of Study)
Description: 1 participant from placebo arm inadvertently received one dose of anifrolumab 1000 milligram (mg).
Arm/Group | Placebo | Anifrolumab 300 mg | Anifrolumab 1000 mg
Serious Adverse Events (participants affected / at risk) | 19/101 | 16/99 | 18/105
Other Adverse Events (participants affected / at risk) | 36/101 | 40/99 | 46/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Anifrolumab 300 mg (N=99) | Anifrolumab 1000 mg (N=105)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 3 (3)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Oedematous kidney (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Anifrolumab 300 mg (N=99) | Anifrolumab 1000 mg (N=105)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (5) | 8 (8)
Bronchitis (Infections and infestations) | 4 (4) | 7 (7) | 9 (11)
Nasopharyngitis (Infections and infestations) | 4 (4) | 12 (15) | 12 (20)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 12 (14) | 11 (20)
Urinary tract infection (Infections and infestations) | 11 (18) | 15 (16) | 7 (12)
Headache (Nervous system disorders) | 13 (21) | 12 (14) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.